CLINICAL TRIAL: NCT01587989
Title: A Multi-center Study of the Safety and Effect on Disease Activity of Tocilizumab (TCZ) in Combination With Methotrexate (MTX) Versus Tocilizumab Monotherapy in Patients With Mild to Moderate Rheumatoid Arthritis, With Inadequate Response to MTX (Defined as DAS 28 < 4,5 and >2,6)
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) With or Without Methotrexate in Patients With Mild to Moderate Rheumatoid Arthritis With an Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML27837; 2011-001863-39 (EudraCT Number)
Record Dates: First submitted 2012-03-12; First posted 2012-04-30 (Estimated); Results first posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A Methotrexate (Active Comparator)
  Interventions: Drug: methotrexate; Drug: tocilizumab [RoActemra/Actemra]
- B Methotrexate Placebo (Experimental)
  Interventions: Drug: methotrexate; Drug: placebo; Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: methotrexate — 15-25 mg orally weekly, Weeks 1-12
Drug: methotrexate — 15-25 mg orally weekly, Weeks 13-24
  Arms: A Methotrexate
Drug: placebo — methotrexate placebo orally weekly, Weeks 13-24
  Arms: B Methotrexate Placebo
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg iv every 4 weeks, 24 weeks

SUMMARY:
This multicenter study with a randomized, double-blind, parallel-group phase will evaluate the safety and efficacy of RoActemra/Actemra (tocilizumab) in combination with methotrexate versus RoActemra/Actemra monotherapy in patients with mild to moderate rheumatoid arthritis, with an inadequate response to methotrexate. Patients will receive RoActemra/Actemra 8 mg/kg intravenously every 4 weeks plus oral methotrexate 15-25 mg weekly for 12 weeks. Patients with a good/moderate EULAR response will then be randomized to receive either RoActemra/Actemra plus methotrexate or RoActemra/Actemra plus placebo for the following 12 weeks. Anticipated time on study treatment is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Rheumatoid arthritis of >/= 1 year duration
* Mild to moderate disease activity at screening (DAS 28 </= 4.5 and >2.6)
* On methotrexate treatment for at least 12 weeks, at stable oral dose of (10)15 mg to 25 mg/week for at least 6 weeks prior to Day 1
* Body weight </= 150 kg
* Oral corticosteroids must have been at stable dose (maximum 10 mg/day) for at least 25 out of 28 days prior to baseline

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months after baseline
* Rheumatic autoimmune disease other than rheumatoid arthritis
* Functional class IV American College of Rheumatology (ACR) Classification
* Prior history of or current inflammatory joint disease other than rheumatoid arthritis
* Treatment with a biologic agent at any time prior to baseline
* Treatment with traditional DMARDs other than methotrexate within 1 month (for leflunomide 3 months) prior to baseline
* Intraarticular or parenteral corticosteroids within 6 weeks prior to baseline
* Previous treatment with tocilizumab
* Pregnant or lactating women
* Uncontrolled disease states, such as asthma, psoriasis or inflammatory bowel disease where flares are commonly treated with oral or parenteral corticosteroids
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections
* History of or currently active primary or secondary immunodeficiency
* Evidence of active malignant disease, malignancies diagnosed within the previous 5 years
* Active tuberculosis requiring treatment within the previous 3 years
* Positive for HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Austria (9):
  - Graz
  - Graz-Eggenberg
  - Hollabrunn
  - Innsbruck
  - Linz
  - Salzburg
  - Stockerau
  - Vienna
  - Wels

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The screening population consisted of men and women with mild-to-moderate active rheumatoid arthritis (RA). Pre-study methotrexate (MTX) administration for at least 12 weeks. Participants experiencing inadequate response to MTX (Disease Activity Score Based on 28 Joints Count [DAS28] 28 less than [<] 4,5 and greater than [>] 2,6) enrolled.
Groups:
- All Participants: Participants received TCZ 8 milligrams per kilogram (mg/kg), intravenously (IV), every 4 weeks, from Weeks 1-12. Participants also received MTX 15 milligrams per week (mg/week) to 25 mg/week at a stable dose, orally (PO) as tablets, once per week, from Weeks 1-12. Participants also received folic acid, greater than or equal to (≥) 5 mg/week, PO, from Weeks 1-12. Participants also received non-sterioidal anti-inflammatory drugs (NSAIDs) and oral corticosteroids (less than or equal to [≤] 10 milligrams per day [mg/day] prednisone or equivalent) according to the standard of care of the treatment site from Weeks 1-12. At Week 12 participants who had achieved a good or moderate European League Against Rheumatism (EULAR) response were randomized to receive TCZ plus (+) continued MTX treatment or TCZ + placebo. Participants without a good or moderate EULAR response were excluded from the study and treated according to the standard of care of the treatment site.
- Group A: TCZ + MTX: During a 12-week run-in period, all participants received TCZ 8 mg/kg, IV, every 4 weeks, from Weeks 1-12. Participants also received MTX 15-25 mg/week at a stable dose, PO as tablets, once per week, from Weeks 1-24. At Week 12, participants who had achieved a good or moderate EULAR response were randomized to receive MTX at the same dose they received from Weeks 1-12, PO as tablets, once per week, from Weeks 12-24. Participants also received TCZ 8 mg/kg, IV, every 4 weeks, from Weeks 12-24. Participants also received NSAIDs and oral corticosteroids (≤ 10 mg/day prednisone or equivalent) according to the standard of care of the treatment site from Weeks 1-24. Participants also received folic acid, ≥ 5 mg/week, PO, from Weeks 1-24.
- Group B: TCZ + Placebo: During a 12-week run-in period, all participants received TCZ 8 mg/kg, IV, every 4 weeks, from Weeks 1-12. Participants also received MTX 15-25 mg/week at a stable dose, PO as tablets, once per week, from Weeks 1-12. At Week 12, participants who had achieved a good or moderate EULAR response were randomized to receive placebo, PO as tablets, once per week, from Weeks 12-24. Participants also received TCZ 8 mg/kg, IV, every 4 weeks, from Weeks 12-24. Participants also received NSAIDs and oral corticosteroids (≤ 10 mg/day prednisone or equivalent) according to the standard of care of the treatment site from Day 1 through Week 24. Participants also received folic acid, ≥ 5 mg/week, PO, from Weeks 1-24.
Period: 12-Week Open-Label Run-In Period
Arm/Group | All Participants | Group A: TCZ + MTX | Group B: TCZ + Placebo
Started | 77 | 0 | 0
Completed | 65 | 0 | 0
Not Completed | 12 | 0 | 0
Not completed — Physician Decision | 7 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — No EULAR Response | 4 | 0 | 0
Period: Randomized Study Treatment
Arm/Group | All Participants | Group A: TCZ + MTX | Group B: TCZ + Placebo
Started | 0 | 32 | 33
Completed | 0 | 30 | 32
Not Completed | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Screening failure | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population: all randomized participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: TCZ + MTX | Group B: TCZ + Placebo | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.78 (11.88) | 57.15 (10.83) | 57.46 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Week 12 (Randomization) to Week 24 in DAS28
Description: The DAS28 is a combined index for measuring disease activity in rheumatoid arthritis (RA). The index includes swollen joint counts (SJC) and tender joint counts (TJC), both scored 0-28 (higher scores indicate higher disease activity), as well as acute phase response (APR) determined as erythrocyte sedimentation rate (ESR), and general health (GH), both scored 1-100 (higher scores indicate higher disease activity). DAS28 was calculated according to the following formula: DAS28 equals (=) [0.56 multiplied by (*) the square root (√) of TJC] plus (+) [0.28 * √ of SJC] + (0.70 * the natural logarithm (ln) ESR in millimeters per hour (mm/h)] + [0.014 * GH in mm visual analogue assessment (VAS)]. A negative change from randomization indicated improvement.
Time Frame: Weeks 12 and 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A: TCZ + MTX | Group B: TCZ + Placebo
Number analyzed (Participants) | 32 | 33
score on a scale | 0.17 (0.83) | -0.16 (1.13)
Statistical Analysis 1: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Test type: Superiority or Other; p = 0.188, t-test, 2 sided; Mean Difference (Final Values) = 0.327, 95% CI 2-sided [-0.165 to 0.820]
Statistical Analysis 2: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; At Week 12; Test type: Superiority or Other; p = 0.015, ANCOVA
Statistical Analysis 3: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Adjusted change in DAS28 score from Weeks 12-24; Test type: Superiority or Other; p = 0.304, ANCOVA

2. Secondary Outcome: Percentage of Participants With DAS28 Remission at Week 24
Description: The DAS28 is a combined index for measuring disease activity in RA. The index includes SJC and TJC, both scored 0-28 (higher scores indicate higher disease activity, as well as APR determined as ESR, and GH, both scored 1-100 (higher scores indicate higher disease activity). DAS28 was calculated according to the following formula: DAS28 = 0.56 * √ of TJC + 0.28 * √ of SJC + 0.70 * ln ESR mm/hr + 0.014 * GH in mm VAS. DAS28 < 2.6 = remission.
Time Frame: Week 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Group A: TCZ + MTX | Group B: TCZ + Placebo
Number analyzed (Participants) | 32 | 33
percentage of participants | 81.25 | 87.50
Statistical Analysis 1: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Test type: Superiority or Other; p = 0.732, Fisher Exact

3. Secondary Outcome: vPercentage of Participants With Clinical Disease Activity Index (CDAI) Remission at Week 24
Description: The CDAI is a combined index for measuring disease activity in RA. CDAI is the sum of TJC and SJC, both scored 0-28 (higher scores indicate higher disease activity), as well as patient global assessment (PGA) and evaluator global assessment (EGA) of disease activity, both scored 0 to 10 centimeter (cm) as assessed by VAS. CDAI was calculated according to the following formula: CDAI = SJC + TJC + PGA + EGA. CDAI < 2.8 = remission.
Time Frame: Week 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Group A: TCZ + MTX | Group B: TCZ + Placebo
Number analyzed (Participants) | 32 | 33
percentage of participants | 34.38 | 53.13
Statistical Analysis 1: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Test type: Superiority or Other; p = 0.207, Fisher Exact

4. Secondary Outcome: Percentage of Participants With Simplified Disease Activity Index (SDAI) Remission at Week 24
Description: The SDAI is a combined index for measuring disease activity in RA. SDAI is the sum of TJC and SJC, both scored 0-28 (higher scores indicate higher disease activity), PGA and EGA of disease activity, both scored 0 to 10 cm as assessed by VAS, and C-reactive protein level (CRP) in milligrams per deciliter (mg/dL) where normal < 1 mg/dL. CDAI was calculated according to the following formula: SDAI = TJC + SJC + PGA + EGA + CRP. SDAI < 3.3 = remission.
Time Frame: Week 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Group A: TCZ + MTX | Group B: TCZ + Placebo
Number analyzed (Participants) | 32 | 33
percentage of participants | 40.63 | 53.13
Statistical Analysis 1: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Test type: Superiority or Other; p = 0.453, Fisher Exact

5. Secondary Outcome: Percentage of Participants With Rheumatoid Arthritis Disease Activity Index-5 (RADAI-5) Remission at Week 24
Description: The RADAI-5 is a combined index for measuring disease activity in RA. RADAI-5 is comprised of the following 5 questions: how active was your arthritis the last 6 months? (0 = completely inactive to 10 = extremely active); how active is your arthritis today with respect to joint tenderness and swelling? (0 = completely inactive to 10 = extremely active); how severe is your arthritis pain today? (0 = no pain to 10 = unbearable pain); how would you describe your general health today? (0 = very good to 10 = very bad); and did you experience joint (hand) stiffness on awakening yesterday morning? If yes, how long did this stiffness last? (0 = no stiffness to 10 = stiffness the whole day). RADAI was calculated according to the following formula: [question (Q) 1 + Q2 + Q3 + Q4 + Q5]/5. RADAI-5 from 0-1.4 = remission.
Time Frame: Week 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Group A: TCZ + MTX | Group B: TCZ + Placebo
Number analyzed (Participants) | 32 | 33
percentage of participants | 32.26 | 54.55
Statistical Analysis 1: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Test type: Superiority or Other; p = 0.084, Fisher Exact

6. Secondary Outcome: Change From Week 12 (Randomization) to Week 24 in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score
Description: HAQ-DI scores were obtained by scoring participants' responses to a 20-item questionnaire. HAQ-DQ evaluated 8 domains of health: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities from a range of 0 (without any difficulty) to 3 (unable to do). The sum of scores was divided by the number of domains for a total score of 0 (best) to 3 (worst). A negative change from randomization indicated improvement.
Time Frame: Weeks 12 and 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A: TCZ + MTX | Group B: TCZ + Placebo
Number analyzed (Participants) | 32 | 33
score on a scale | 0.04 (0.28) | -0.06 (0.40)
Statistical Analysis 1: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Test type: Superiority or Other; p = 0.842, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change From Week 12 (Randomization) to Week 24 in Short Form-36 Health Survey (SF-36) Score
Description: SF-36 scores were obtained by scoring participants' responses to a 36-item questionnaire. SF-36 evaluated 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health from a range of 1 (better) to 5 (worst). The score for each section was an average of the individual question scores, which were scaled 0-100 (100=highest level of functioning). These 8 aspects were summarized as physical and mental component scores. A negative change from randomization indicated improvement.
Time Frame: Weeks 12 and 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A: TCZ + MTX | Group B: TCZ + Placebo
Number analyzed (Participants) | 32 | 33
score on a scale
  Physical standardized value | 0.89 (10.48) | 0.75 (10.08)
  Mental standardized value | -5.41 (9.24) | -1.69 (9.20)
Statistical Analysis 1: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Physical standardized value; Test type: Superiority or Other; p = 0.417, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Mental standardized value; Test type: Superiority or Other; p = 0.112, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change From Week 12 (Randomization) to Week 24 in Visual Analog Scales (VAS) Scores
Description: VAS scores were obtained by scoring participants' disease activity as assessed on a 0-100 millimeter (mm) horizontal visual scale. The left-hand extreme of the line = 0 mm (no disease activity = symptom-free and no arthritis symptoms), and the right-hand extreme of the line = 100 mm (maximum disease activity). A negative change from randomization indicated improvement.
Time Frame: Weeks 12 and 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A: TCZ + MTX | Group B: TCZ + Placebo
Number analyzed (Participants) | 32 | 33
score on a scale
  Fatigue | 1.91 (17.16) | -1.88 (17.49)
  Pain | 1.09 (18.48) | -2.88 (22.04)
Statistical Analysis 1: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Fatigue; Test type: Superiority or Other; p = 0.655, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Pain; Test type: Superiority or Other; p = 0.839, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Participant Satisfaction With Treatment as Assessed by Treatment Satisfaction Questionnaire for Medication (TSQM) Score
Description: TSQM scores were obtained by scoring participants' responses to a 14-item questionnaire. TSQM evaluated 4 aspects of treatment satisfaction: effectiveness, side effects, convenience, and global satisfaction from a range of 0 to 100 percent (%), with 100% being the best possible result.
Time Frame: Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A: TCZ + MTX | Group B: TCZ + Placebo
Number analyzed (Participants) | 32 | 33
score on a scale
  Effectiveness | 72.41 (34.85) | 82.49 (24.14)
  Side-effects | 94.15 (19.16) | 94.89 (14.70)
  Convenience | 85.48 (21.97) | 86.03 (15.60)
  Global satisfaction | 86.64 (21.09) | 86.36 (13.53)
Statistical Analysis 1: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Effectiveness; Test type: Superiority or Other; p = 0.580, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Side-effects; Test type: Superiority or Other; p = 0.975, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Convenience; Test type: Superiority or Other; p = 0.421, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group A: TCZ + MTX vs Group B: TCZ + Placebo; Global satisfaction; Test type: Superiority or Other; p = 0.277, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from Weeks 12-24.
Description: All randomized participants who received at least 1 dose of treatment were included in the safety analysis.
Arm/Group | Group A: TCZ + MTX | Group B: TCZ + Placebo
Serious Adverse Events (participants affected / at risk) | 2/32 | 5/33
Other Adverse Events (participants affected / at risk) | 14/32 | 12/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: TCZ + MTX (N=32) | Group B: TCZ + Placebo (N=33)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: TCZ + MTX (N=32) | Group B: TCZ + Placebo (N=33)
Leukopenia (Blood and lymphatic system disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 3 | 5
Nasopharyngitis (Infections and infestations) | 5 | 1
Oral herpes (Infections and infestations) | 1 | 5
Alanine aminotransferase increased (Investigations) | 4 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.